CLINICAL TRIAL: NCT01604226
Title: Predicting Bispectral Index Values by Estimated Effect-site Concentration of Propofol and Remifentanil Displayed on the Target-centered Infusion Pump
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin M. Lee, Professor, Samsung Medical Center
Other Study IDs: 2012-04-094
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: General Anesthesia; Total Intravenous Anesthesia; Bispectral Index Monitoring
Keywords: total intravenous anesthesia; Bispectral index monitoring; propofol; remifentanil

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gynecologic surgery group: Those undergoing gynecologic laparoscopic surgery with TIVA
- Urologic surgery group: Those undergoing urologic surgery with TIVA

SUMMARY:
The BIS is influenced by multiple parameters, such as age,gender, body weight, height, muscle relaxants, hepatic function, co-administered drugs, surgical stimulation, but is thought to be influenced mainly by propofol and remifentanil infusion dose. As such, the investigators postulate that the BIS value could be predicted by the estimated effects-site concentration of propofol and remifentanil, and try to establish a multiple linear regression model for predicting BIS value.

DETAILED DESCRIPTION:
Total intravenous anesthesia is commonly performed with propofol and remifentanil now-a-days. The combination of these two drugs can achieve the rapid loss of consciousness and analgesia,as the onset and recovery time of these two drugs are very fast within one to three minutes. However, the problem of intraoperative awareness necessitate the monitoring of anesthetic depth, which is commonly performed with Bispectral index (BIS). BIS is a display of number from zero to one hundred which quantify the degree of sedation and hypnosis by anesthetics by analyzing the electroencephalogram. However, it is limited in neurosurgery in which the surgical field is near the forehead where the BIS probe is attached. Furthermore, it is also limited in surgery with prone position. The BIS is influenced by multiple parameters, such as age,gender, body weight, height, muscle relaxants, hepatic function, co-administered drugs, surgical stimulation, but is thought to be influenced mainly by propofol and remifentanil infusion dose. As such, we postulate that the BIS value could be predicted by the estimated effects-site concentration of propofol and remifentanil, and try to establish a multiple linear regression model for predicting BIS value.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing gynecologic or urologic surgery with general anesthesia with total intravenous anesthesia
* Adult patients with more than 20 yrs.
* American Society of Anesthesiologists Class I or II.

Exclusion Criteria:

* Those with unstable hemodynamics
* Those who can not undergo Bispectral index monitoring
* Those with previous history of stroke

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those undergoing gynecologic or urologic surgery with general anesthesia with total intravenous anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Bispectral index value | every 10 min after anesthetic induction
  Bispectral index value after anesthetic induction every 10 minutes interval until the end of surgery

SECONDARY OUTCOMES:
Propofol concentration | every 10 min after anesthetic inducton
  estimated propofol effect-site concentration displayed in target-centered infusion pump every 10 minutes interval
Remifentanil concentration | every 10 minutes after anesthetic induction
  estimated remifentanil effect-site concentration displayed in target-centered infusion pump every 10 minutes interval

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin M. Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea